CLINICAL TRIAL: NCT01174173
Title: Effects of Ranolazine in Patients With Angina Due to Right Ventricular Ischemia in Pulmonary Arterial Hypertension
Brief Title: Ranolazine and Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Sanjiv Shah, Principal Invesitgator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00030314
Record Dates: First submitted 2010-07-23; First posted 2010-08-03 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Angina; Pulmonary Arterial Hypertension
Keywords: Angina; Right Ventricular Ischemia; Pulmonary Arterial Hypertension; Pulmonary Hypertension
MeSH Terms: conditions — Angina Pectoris; Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranolazine (Experimental): 1000 mg PO BID
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — ranolazine 1000 mg PO BID for 3 months
  Other Names: Ranexa

SUMMARY:
The purpose of the study is to determine if the medication, ranolazine (study drug), can help improve blood flow to your heart, increase your exercise capacity and improve your quality of life (QOL). For this study, you will be asked to perform several tests in order to determine if your heart function, exercise capacity, chest pain and QOL have improved after 3 months of treatment with ranolazine. Ranolazine is approved by the U.S. Food and Drug Administration (FDA) for the treatment of angina.

DETAILED DESCRIPTION:
This study is looking to enroll patients with pulmonary hypertension (PH). PH is abnormally high blood pressure in the arteries of the lungs. It makes the right side of the heart need to work harder than normal and is usually caused by a narrowing of the small arteries of the lung. This narrowing makes it harder for the right side of the heart to circulate the blood to the lungs. Over time, the right side of the heart may become enlarged and symptoms (such as angina [chest pain] shortness of breath, fatigue, edema) begin to appear.

Ranolazine is a safe, well-tolerated, and FDA-approved medication for the treatment of chronic stable angina. Ranolazine may potentially improve blood flow to the right ventricle (RV), thereby relieving angina while simultaneously improving RV performance and contractility. This latter effect may increase stroke volume and cardiac output which could translate into benefits in exercise capacity and improved quality of life.

The purpose of this single center, non-randomized, prospective pilot study is to investigate the effects of 3 months treatment with ranolazine on pulmonary artery hemodynamics, exercise capacity and quality of life in patients with PAH and symptoms of angina or angina equivalent.

ELIGIBILITY:
Inclusion criteria:

1. World Health Organization (WHO) Group 1 PAH, defined as a pulmonary hypertension with mean pulmonary artery pressure > 25 mmHg, pulmonary capillary wedge pressure < 15 mmHg, and pulmonary vascular resistance > 3 Wood units.
2. Right ventricular dysfunction, defined as RV fractional area change < 32% or RV tricuspid annular plane systolic excursion (TAPSE) < 15 mm.
3. Symptoms of angina or angina equivalent (exertional dyspnea, exertional epigastric pain, exertional nausea).
4. New York Heart Association functional class II or III symptoms.
5. Stable doses of pulmonary vasodilators (prostacyclins, endothelin receptor antagonists, phosphodiesterase inhibitors), with no new therapy initiation or dose escalation > 50% in the 4 weeks prior to randomization.
6. Age 18-80 years.

Exclusion criteria:

1. Acute coronary syndrome or coronary revascularization within the prior 3 months.
2. Patients with unstable angina.
3. Patients with Class IV congestive heart failure.
4. Planned revascularization, pacemaker or defibrillator placement during the study period.
5. Changes in antianginal medical therapy likely to occur during the study period.
6. Corrected QT interval measurement >500 ms.
7. Patients with pre-existing QT prolongation (including congenital long QT syndrome) or receiving other QT prolonging drugs (including Class Ia-e.g., quinidine, Class III-e.g., dofetilide, sotalol, antiarrhythmics; antipsychotics (e.g., thioridazine, ziprasidone), or known history of complex ventricular arrhythmias requiring antiarrhythmic medications or ICD implantation.
8. Patients with known history of hepatic dysfunction.
9. Current use of strong CYP3A inhibitors, including ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, saquinavir and diltizaem.
10. Patients with pacemakers, cochlear implants, aneurysm clips, who have worked with metal.
11. Patients with metallic hardware, implants, or prostheses will consult with the radiologist/cardiologist prior to the study.
12. Patients with severe or end stage renal disease (an estimated GFR < 30 mL/min/1.73 m).
13. Women who are pregnant or lactating
14. Any contraindications for the use of a right heart catheter including, but not limited to:

    * Pulmonic or tricuspid valve stenosis
    * Prosthetic pulmonic or tricuspid valve
    * Right atrial or ventricular masses
    * Previous pneumonectomy
    * Risk of severe arrhythmias, including left bundle branch block (LBBB)
15. Subjects unable to perform cardiopulmonary exercise testing will be excluded (i.e. extensive musculoskeletal disease)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-06; Primary Completion 2014-01 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Khan SS, Cuttica MJ, Beussink-Nelson L, Kozyleva A, Sanchez C, Mkrdichian H, Selvaraj S, Dematte JE, Lee DC, Shah SJ. Effects of ranolazine on exercise capacity, right ventricular indices, and hemodynamic characteristics in pulmonary arterial hypertension: a pilot study. Pulm Circ. 2015 Sep;5(3):547-56. doi: 10.1086/682427. PMID 26401256
- See also: Bluhm Cardiovascular Institute Clinical Trials Unit research studies — http://www.feinberg.northwestern.edu/ctu/current_research/heart_failure/index.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine
Started | 11
Completed | 10
Not Completed | 1
Not completed — drug-drug interaction | 1

BASELINE CHARACTERISTICS:
Population: We prospectively enrolled 11 patients with WHO Group 1 PAH with mean age was 48±13 years and 73% of patients were women. Nearly half of the study participants were non-white.
Arm/Group | Ranolazine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11
Exercise stress echocardiography with strain [Mean (Standard Deviation); unit: Ejection Fraction (%)] | 63 (5)
Right heart catheterization [Mean (Standard Deviation); unit: Mean pulmonary artery pressure (mm Hg)] | 48 (14)
6-minute walk test [Mean (Standard Deviation); unit: meters] | 383 (60)

OUTCOME MEASURES:

1. Primary Outcome: Improve Angina Symptoms
Description: Assessed as average improvement in WHO Functional Class. The WHO Functional Class score ranges from 1 to 4, with higher scores indicating more impairment
Time Frame: 3 months
Population: Analysis was performed on all participants who completed as average change in WHO Functional class score from baseline to 3 months (Baseline, 3 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranolazine
Number analyzed (Participants) | 8
units on a scale | 1.75 (0.46)
Statistical Analysis 1: Comparison: Ranolazine; Test type: Superiority or Other; p = 0.0013, t-test, 2 sided — A two-sided t-test was performed with p-value < 0.05 was considered statistically significant a priori

2. Primary Outcome: 6-Minute Walk Test
Description: Improve Exercise Capacity measured by 6-Minute Walk Test
Time Frame: 3 Months
Population: Analysis was performed in all participants who completed the study and had a 6-minute walk test at baseline and at the conclusion of the study.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ranolazine
Number analyzed (Participants) | 6
meters | 419 (80)
Statistical Analysis 1: Comparison: Ranolazine; Test type: Superiority or Other; p = 0.09, t-test, 2 sided — A two-sided t-test was performed for change in 6-minute walk test and p-value < 0.05 was considered statistically significant a priori

3. Primary Outcome: Improve Quality of Life
Description: The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The scores are averaged and transformed to a range of 0-100, in which higher scores reflect better health status and was performed at the conclusion of the study.
Time Frame: 3 Months
Population: Analysis was performed on the 8 participants who completed the KCCQ questionnaire at baseline and at the conclusion of the study (month 3)
Measure: Mean (Standard Deviation); unit: KCCQ Summary Score
Arm/Group | Ranolazine
Number analyzed (Participants) | 8
KCCQ Summary Score
  Baseline | 60.3 (19.7)
  Month 3 | 64.2 (17.5)
Statistical Analysis 1: Comparison: Ranolazine; Test type: Superiority or Other; p = 0.37, t-test, 2 sided — A two-sided t-test was performed for difference from baseline and 3-month KCCQ score. A p-value of <0.05 was considered statistically significant a priori

4. Secondary Outcome: RV Perfusion on Cardiac MRI
Description: The majority of patients did not undergo cardiac MRI because it was difficult for the patients to tolerate the imaging study. Therefore, we were not able to assess change in RV perfusion.
Time Frame: 3 months
Groups:
- Ranolazine 1000 mg po Bid: MRI was not analyzable due to inability of patients to undergo MRI due to technical issues
Arm/Group | Ranolazine 1000 mg po Bid
Number analyzed (Participants) | 0

5. Secondary Outcome: Absolute RV Longitudinal Strain
Description: Change in absolute right ventricular (RV) longitudinal strain as assessed by exercise stress echocardiography with speckle-tracking echocardiography at baseline and conclusion of the study. An increase in exercise-induced change in RV longitudinal strain between baseline to conclusion of the study is indicative of improved RV function. If absolute RV longitudinal strain increases with exercise, that is a sign that the RV is working well. If absolute RV longitudinal strain decreases with exercise, that is a sign that the RV is not working well. Therefore, between baseline and conclusion of the study, if exercise-induced change in RV strain increases that means that the RV is working better at the conclusion of the study.
Time Frame: 3 months
Population: Analysis was performed on all participants who completed exercise stress echocardiography at baseline and conclusion of the study (month 3)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Ranolazine
Number analyzed (Participants) | 8
percentage
  Baseline | -1.4 (0.7)
  Month 3 | 1.0 (0.5)
Statistical Analysis 1: Comparison: Ranolazine; Test type: Superiority or Other; p = 0.037, t-test, 2 sided

6. Secondary Outcome: Right Ventricular Hemodynamics
Description: Mean pulmonary artery pressure was assessed invasively by right heart catheterization at the conclusion of the study to estimate right ventricular hemodynamics.
Time Frame: 3 months
Population: Analysis was performed on all participants who completed right heart catheterization at the conclusion of the study
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Ranolazine
Number analyzed (Participants) | 8
mm Hg | 48 (6)
Statistical Analysis 1: Comparison: Ranolazine; Test type: Superiority or Other; p = 0.66, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Ranolazine
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=11)
Inpatient hospitalization (Nervous system disorders) | 1 (1) — 1 patient reported symptoms of dizziness, leg weakness, and hand tremors; Because of possibility of an interaction between ranolazine and darifenacin, ranolazine was discontinued, patient withdrawn from the study, and had complete resolution.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=11)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was a small pilot Interventional study to test safety and tolerability of ranolazine in 11 patients with sx WHO Group 1 PAH patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No